CLINICAL TRIAL: NCT06485492
Title: Prospective, Multicenter Design of Clinical Trials to Evaluate the Safety and Efficacy of Aneurysm Embolization Systems for the Treatment of Intracranial Aneurysms, Including Ruptured Aneurysms
Brief Title: Aneurysm Embolization System for Intracranial Aneurysms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu CED Medtech Co., Ltd (Industry)
Responsible Party: Principal Investigator, Jindou Feng, archiater, Jiangsu CED Medtech Co., Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CER-A-AES-01
Record Dates: First submitted 2024-06-17; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Ruptured Cerebral Aneurysm

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, single-group, target-controlled clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Procedure: Implant an aneurysm embolization system

INTERVENTIONS:
Procedure: Implant an aneurysm embolization system — The product uses minimally invasive interventional method to treat intracranial aneurysms approved for application. The study physician selects the appropriate size and/or shape of the aneurysm based on the size and shape of the intracranial arterioma. The aneurysm embolization system device is inserted into the arterioma through a compatible neurovascular microcatheter.

SUMMARY:
The purpose of this clinical study was to evaluate the safety and efficacy of the aneurysm embolization system produced by Jiangsu Changyida Medical Technology Co., Ltd. in patients with intracranial aneurysms (including ruptured aneurysms)

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥18 years old, and ≤75 years old, male or female; (2) There was an unruptured aneurysm or a single ruptured aneurysm requiring treatment, and the Hunt-Hess score was grade I-III; (3) The target aneurysm to be treated must have the following characteristics:

  1. sacculate;
  2. aneurysms located in anterior communicating artery, middle cerebral artery bifurcation aneurysms and basilar artery apex aneurysms;
  3. The diameter of the aneurysm is in accordance with the instruction manual of the aneurysm embolization system for treatment;
  4. Aneurysm diameter from 2mm to 15mm;
  5. Tumor body/neck (D/N) ratio ≥1;
  6. Tumor neck ≥4mm or tumor body/neck (D/N) ratio < 2; (4) The target aneurysm is suitable for aneurysm embolization system treatment; (5) The subject is able to understand the purpose of the study, demonstrates sufficient adherence to the study protocol, and is able and willing to sign the informed consent.

Exclusion Criteria:

* (1) Patients with aneurysms who are not suitable for endovascular therapy; (2) The microcatheter could not reach the target aneurysm of the patient after being shaped, and could not be treated with research instruments; (3) There are risk factors for ischemic stroke, or ischemic symptoms that have occurred within the last 30 days, such as transient ischemic attack, minor stroke, or progressive stroke; (4) The presence of cerebrovascular, cardiovascular or neurological diseases that cause instability of neurological symptoms; (5) mRS≥ 2 before the onset of symptoms or rupture of the aneurysm (if applicable); (6) Patients with intracranial hypertension or other intracranial hematoma within 90 days requiring elective surgery; (7) Patients who are being treated with anticoagulants or who currently have malignant diseases of the blood system, coagulation diseases or hemoglobinopathy; (8) Patients who are allergic to any component of the research instrument, surgical material or drugs used during the operation and cannot be effectively treated; (9) Patients whose life expectancy is less than 2 years due to other diseases or conditions (other than intracranial aneurysms); (10) Patients with mental disorders; (11) Women who are pregnant or breastfeeding, or who have a birth plan in the next 3 months; (12) Patients who are participating in any other drug or medical device clinical trial, or who may participate in any other drug or medical device clinical trial after enrollment in this clinical trial; (13) The investigator determines that there are other conditions that are not suitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Adequate embolization rate at 1 year follow-up. | 1year
  Full embolization means that the aneurysm is completely occluded or only the neck remains.

IPD SHARING:
Plan to Share IPD: No